CLINICAL TRIAL: NCT02819284
Title: A Phase 3, Double-Masked, Randomized, Controlled Study of KPI-121 0.25% Ophthalmic Suspension Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: Safety and Efficacy of KPI-121 Compared to Placebo in Subjects With Dry Eye Disease
Acronym: STRIDE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-007
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
Keywords: Ocular Discomfort; Pain; Corticosteroid; Hyperemia; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Pain; Hyperemia | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KPI-121 0.25% Ophthalmic Suspension (Active Comparator)
  Interventions: Drug: KPI-121 0.25% Ophthalmic Suspension
- Vehicle of KPI-121 0.25% Ophthalmic Suspension (Placebo Comparator)
  Interventions: Drug: Vehicle of KPI-121 0.25% Ophthalmic Suspension

INTERVENTIONS:
Drug: KPI-121 0.25% Ophthalmic Suspension
  Other Names: Loteprednol etabonate
  Arms: KPI-121 0.25% Ophthalmic Suspension
Drug: Vehicle of KPI-121 0.25% Ophthalmic Suspension
  Other Names: Placebo
  Arms: Vehicle of KPI-121 0.25% Ophthalmic Suspension

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of KPI-121 0.25% ophthalmic suspension compared to vehicle (placebo) in subjects who have a documented clinical diagnosis of dry eye disease. The product will be studied over 14 days, with 1-2 drops instilled in each eye four times daily (QID).

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the safety and efficacy of KPI-121 0.25% ophthalmic suspension versus vehicle in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented clinical diagnosis of dry eye disease in both eyes

Exclusion Criteria:

* Known hypersensitivity or contraindication to the investigational product(s) or components
* History of glaucoma, IOP>21 mmHg at the screening or randomization visits, or being treated for glaucoma in either eye.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within 30 days prior to screening.
* In the opinion of the Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - UAB School of Optometry, Birmingham, Alabama
  - Arizona Eye Center, Chandler, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Sall Research Medical Center, Artesia, California
  - Milton M. Hom, OD, FAAO, Azusa, California
  - Family Eye Care Center, Campbell, California
  - Orange County Ophthalmology, Garden Grove, California
  - Lugene Eye Institute, Glendale, California
  - The Gavin Herbert Eye Institute, Irvine, California
  - Macy Eye Center, Los Angeles, California
  - Advanced Vision Care, Los Angeles, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Arch Health Partners, Poway, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc, Redding, California
  - West Coast Eye Care Associates, San Diego, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Michael K Tran, M.D., Inc., Westminster, California
  - Hernando Eye Institute, Brooksville, Florida
  - Central Florida Eye Associates, Lakeland, Florida
  - Shettle Eye Research, Inc, Largo, Florida
  - International Eye Associates PA, Ormond Beach, Florida
  - Perez Eye Center/International Research Center, Tampa, Florida
  - Eye Care Centers Management, Inc. (Clayton Eye Center), Morrow, Georgia
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Koffler Vision Group, Lexington, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Taustine Eye Center, Louisville, Kentucky
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Minnesota Eye Consultants, PA, Bloomington, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Comprehensive Eye Care, Ltd. / Vision Research Institute, LLC, Washington, Missouri
  - Abrams Eye Institute, Las Vegas, Nevada
  - Raymond Fong, MDPC, New York, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - James D Branch MD, Winston-Salem, North Carolina
  - Comprehensive Eye Care of Central Ohio, Westerville, Ohio
  - Drs. Fine, Hoffman & Sims, LLC, Eugene, Oregon
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania
  - Chattanooga Eye Institute, P.C., Chattanooga, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Toyos Clinic, Nashville, Tennessee
  - Texan Eye, PA / Keystone Research, Ltd, Austin, Texas
  - The Cataract and Glaucoma Center, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Advanced Laser Vision & Surgical Institute, Intouch Clinical Research Center, Houston, Texas
  - Whitsett Vision Group, Houston, Texas
  - The Ocular Surface Institute (TOSI), University of Houston, Houston, Texas
  - Brazosport Eye Institute, Lake Jackson, Texas
  - Kozlovsky Delay & Winter Eye Consultants, LLC, San Antonio, Texas
  - Hoopes Vision, Draper, Utah
  - Virginia Eye Consultants, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
  - Regional Eye Associates, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 909 subjects were randomized, 4 of which were not included in any analysis population as agreed upon with the FDA. 3 individuals had participated in more than one study therefore the data for their second-participation were not included and 1 individual did not receive treatment.
Groups:
- KPI-121 0.25% Ophthalmic Suspension: Participants randomized to KPI-121 0.25% Ophthalmic Suspension
- Vehicle of KPI-121 0.25% Ophthalmic Suspension: Participants randomized to Vehicle of KPI-121 0.25% Ophthalmic Suspension
Period: Overall Study
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Started | 452 | 453
Completed | 447 | 448
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension | Total
Number analyzed (Participants) | 452 | 453 | 905
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (14.48) | 59.3 (15.01) | 59.2 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332 | 354 | 686
  Male | 120 | 99 | 219
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 39 | 35 | 74
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 58 | 54 | 112
  White | 345 | 352 | 697
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 452 | 453 | 905

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline/Visit 2 (Day 1) in Bulbar Conjunctival Hyperemia at Visit 4 (Day 15)
Description: Comparison of mean change from baseline for bulbar conjunctival hyperemia in the study eye between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-4 grading scale. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: Intent to Treat population minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 446 | 447
score on a scale | -0.3812 (0.60560) | -0.2371 (0.62256)

2. Primary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Severity at Visit 4 (Day 15)
Description: Comparison of mean ocular discomfort between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 445 | 444
score on a scale | -11.14 (19.901) | -9.24 (17.002)

3. Secondary Outcome: Proportion of Subjects With ≥ 1 Unit Improvement From Baseline/Visit 2 (Day 1) in Bulbar Conjunctival Hyperemia Worst Region at Visit 4 (Day 15)
Description: Proportion of subjects with ≥1 improvement from baseline in conjunctival hyperemia scores in the study eye. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 446 | 447
Participants | 171 | 127

4. Secondary Outcome: Change From Baseline/ Visit 2 (Day 1) in Ocular Discomfort Severity Scores at Visit 3 (Day 8)
Description: Comparison of ocular discomfort scores between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse using 3-day mean scores.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 3 (Day 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 449 | 451
score on a scale | -6.92 (15.541) | -4.86 (14.911)

5. Secondary Outcome: Change From Baseline/Week 2 (Day 1) in Ocular Discomfort Scores to Day 4
Description: as for outcome 2
Time Frame: Baseline/Visit 2 (Day 1) - Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 447 | 449
score on a scale | -5.09 (14.523) | -4.10 (14.894)

6. Secondary Outcome: Change From Baseline/Week 2 (Day 1) in Ocular Discomfort Severity at Visit 4 (Day 15) in a Subgroup
Description: Comparison of mean ocular discomfort between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse, in a sub-group of participants with more severe ocular discomfort at baseline, using 3 day means.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: Sub-group of Intent to Treat population with more severe ocular discomfort minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 254 | 257
score on a scale | -12.45 (20.352) | -9.45 (17.489)

7. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Severity Scores at Day 3 (Diary)
Description: Comparison of mean ocular discomfort severity between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Baseline/Visit 2 (Day 1) - Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 451 | 449
score on a scale | -3.28 (13.697) | -3.15 (14.126)

8. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Eye Dryness Scores at Visit 4 (Day 15)
Description: Comparison of mean eye dryness between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 447 | 445
score on a scale | -14.0 (22.78) | -11.5 (20.53)

9. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Eye Dryness Scores at Visit 3 (Day 8)
Description: as for outcome 8
Time Frame: Baseline/Visit 2 (Day 1) - Visit 3 (Day 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 442 | 447
score on a scale | -9.6 (18.66) | -8.0 (18.94)

10. Secondary Outcome: Ocular Discomfort Severity Scores on Day 2 (Diary) Minus Baseline/Visit 2 (Day 1)
Description: as for outcome 2
Time Frame: Baseline/Visit 2 (Day 1) - Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 451 | 447
score on a scale | -2.33 (13.707) | -2.43 (13.364)

11. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Frequency Scores at Visit 4 (Day 15)
Description: Comparison of mean ocular discomfort frequency between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 445 | 444
score on a scale | -10.20 (20.722) | -8.38 (17.974)

12. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Subject-rated Ocular Discomfort Frequency Scores at Visit 3 (Day 8)
Description: as for outcome 11
Time Frame: Baseline/Visit 2 (Day 1) - Visit 3 (Day 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 449 | 451
score on a scale | -5.96 (16.133) | -4.42 (16.133)

13. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Inferior Corneal Fluorescein Staining Score at Visit 4 (Day 15)
Description: Comparison of mean corneal fluorescein staining in the study eye between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using methods developed by the National Eye Institute (NEI) Dry Eye Workshop in evaluating 5 regions of the cornea (superior, inferior, nasal, temporal and central) using a 0-3 grading scale, where 0 = no visible staining, 1 = Mild, 2 = moderate and 3 = severe.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 448 | 448
score on a scale | -0.6 (0.86) | -0.5 (0.83)

14. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Nasal Corneal Fluorescein Staining Score at Visit 4 (Day 15)
Description: Comparison of mean nasal corneal fluorescein staining in the study eye between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using methods developed by the National Eye Institute (NEI) Dry Eye Workshop in evaluating 5 regions of the cornea (superior, inferior, nasal, temporal and central) using a 0-3 grading scale, where 0 = no visible staining, 1 = Mild, 2 = moderate and 3 = severe.
Time Frame: Baseline/Visit 2 (Day 1) - Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 448 | 448
score on a scale | -0.6 (0.86) | -0.4 (0.83)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 2 (Day 1) until they exited the study at Visit 4 (Day 15).
Description: Both treatment-related and non-treatment-related adverse events are reported here.
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/452 | 0/453
Serious Adverse Events (participants affected / at risk) | 3/452 | 0/453
Other Adverse Events (participants affected / at risk) | 57/452 | 44/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=452) | Vehicle of KPI-121 0.25% Ophthalmic Suspension (N=453)
diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=452) | Vehicle of KPI-121 0.25% Ophthalmic Suspension (N=453)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Eye pruritus (Eye disorders) | 3 | 4
Conjunctival hyperaemia (Eye disorders) | 2 | 3
Eye irritation (Eye disorders) | 2 | 4
Eye pain (Eye disorders) | 2 | 3
Conjunctival haemorrhage (Eye disorders) | 1 | 2
Conjunctival oedema (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Eyelid pruritus (Eye disorders) | 1 | 0
Iritis (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 6
Vision acuity reduced (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Corneal infiltrates (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastroesophogeal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Instillation site pain (General disorders) | 26 | 20
Chest pain (General disorders) | 1 | 0
Instillation site discharge (General disorders) | 1 | 0
Instillation site irritation (General disorders) | 1 | 0
Instillation site pruritus (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Body tinea (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Vaginal infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 2
Ophthalmoplegic migraine (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between the Principal Investigator and the Sponsor restricts the PI's rights to discuss or publish trial results until after the first to occur of the following:

(a) publication of such multi-center clinical trial results; (b) notification by sponsor that such a multi-center clinical trial submission is no longer planned; or ( c) the eighteen ( 18) month anniversary of the completion, abandonment or termination of such multi-center clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02819284/Prot_SAP_000.pdf